CLINICAL TRIAL: NCT03482557
Title: Contrast Enhanced Spectral Mammography vs. MRI for Breast Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: GE Healthcare (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Olga Brook, Vice-Chair of Research, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 17-689
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; screening; breast MRI; contrast enhanced spectral mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Contrast-Enhanced Spectral Mammography (Experimental): Each enrolled participant will receive a CESM either at the time of screening or following screening, for a screen detected finding. If patient has a biopsy for a finding, the CESM must be performed prior to biopsy.
  Interventions: Device: CESM
- Breast MRI (Experimental): Each enrolled participant will receive an MRI exam either at the time of screening or following screening, for a screen detected finding. If patient has a biopsy for a finding, the MRI must be performed prior to biopsy.
  Interventions: Device: MRI

INTERVENTIONS:
Device: CESM — Contrast enhanced mammography is a new type of mammogram. It uses contrast material combined with the mammogram to highlight areas that might be breast cancer and that could be missed on the mammogram alone
  Other Names: Contrast Enhanced Spectral Mammography
  Arms: Contrast-Enhanced Spectral Mammography
Device: MRI — MRI uses magnets to create a detailed image of the tissues and bones inside of the body
  Other Names: Magnetic Resonance Imaging
  Arms: Breast MRI

SUMMARY:
This research study is evaluating whether contrast enhanced mammography can be used as an alternative to breast Magnetic Resonance Imaging (MRI) for cancer screening

DETAILED DESCRIPTION:
Mammography is the main way to help find breast cancers early so they can be treated. Unfortunately, mammography does not work as well in women who have dense breast tissue or who are at high-risk for breast cancer. In these women, breast MRI is also used to help find breast cancers.

Contrast enhanced mammography is a new type of mammogram. It uses contrast material combined with the mammogram to highlight areas that might be breast cancer and that could be missed on the mammogram alone. This is similar to breast MRI.

For this study, participants who had both CEM and MRI evaluating a finding that initiated from a screening exam will be included. Radiologists will compare the images to see if the contrast enhanced mammograms and the breast MRI find the same number of breast cancers. If the investigators find they perform similarly, then contrast mammography may be used to aid in breast cancer screening in the future.

ELIGIBILITY:
Inclusion Criteria:

* CESM and MRI exam performed within 3 months of one another.
* CESM and breast MRI exams must be performed as part of imaging work-up based on a screening exam of any type (mammography, tomosynthesis, ultrasound, and MRI)
* CESM studies will include at least four low energy and four recombined images (LCC, LMLO, RCC, RMLO).
* MRI exams will include at least fluid sensitive sequence, multi-phase T1-weighted

Exclusion Criteria:

* Imaging sets with implants.
* Imaging sets in which a biopsy or surgical intervention was performed since the most recent screening exam, prior to acquisition of the study MRI or CESM.
* Imaging sets in which a biopsy was recommended, but biopsy was not performed and 2 year imaging follow-up is not available

Ages: 30 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Brook, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 132
Pre-assignment Details: 132 patients were included in the reader study. 42 patients had imaging acquired as part of clinical trial NCT02275871, 78 as part of clinical trial NCT03482557, and 12 as part of clinical care.
Groups:
- Screening CESM and MRI: Each enrolled participant will receive both a CESM and MRI exam either at the time of screening or following screening, for a screen detected finding. If patient has a biopsy for a finding, the CEM and MRI must be performed prior to biopsy.
Period: Overall Study
Arm/Group | Screening CESM and MRI
Started | 132
Completed | 132
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Screening CESM and Breast MRI: Each enrolled participant will receive both a CESM and MRI exam either at the time of screening or following screening, for a screen detected finding. If patient has a biopsy for a finding, the CEM and MRI must be performed prior to biopsy.
Arm/Group | Screening CESM and Breast MRI
Number analyzed (Participants) | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 116
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 54 [30 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 132

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Cancer Detection Rates of CESM Compared With Breast MRI for Breast Cancer Screening
Description: We will determine whether CESM is non-inferior to breast MRI for breast cancer detection by comparing cancer detection rates on both studies using a multi-case multi-reader study model.
Time Frame: 2 years
Population: Images from 78 patients were included from prospective recruitment, images from 42 patients from prior research (NCT02275871), and images from 12 patients from clinical care.
Measure: Number (95% Confidence Interval); unit: Probability of malignancy
Groups:
- Cancers Identified With CESM; Cancers Identified With Screening MRI: Recruited patient images were added to other patient images who had both CEM and MRI before biopsy. The images were included in a reader study evaluating diagnostic accuracy of CEM vs MRI
Arm/Group | Cancers Identified With CESM | Cancers Identified With Screening MRI
Number analyzed (Participants) | 132 | 132
Probability of malignancy | 0.91 [.885 to 0.926] | .91 [0.894 to 0.925]

2. Secondary Outcome: Area Under the Curve for Cancer Detection Rates of CESM Compared With Abbreviated Breast MRI for Breast Cancer Screening
Description: Radiologist readers evaluated CEM and abbreviated MRI in 132 patients, some who had cancer and some who did not. The area under the curve was determine for each reader for each exam type.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of malignancy
Groups:
- CESM; Screening Abbreviated MRI: Recruited patient images were added to other patient images who had both CEM and MRI before biopsy. The images were included in a reader study evaluating diagnostic accuracy of CEM vs abbreviated MRI
Arm/Group | CESM | Screening Abbreviated MRI
Number analyzed (Participants) | 132 | 132
Probability of malignancy | .906 [.885 to 0.926] | .894 [.859 to .929]

3. Secondary Outcome: Area Under the Curve for Cancer Detection Rates of CESM Compared With Conventional 2d Mammography for Breast Cancer Screening
Description: We will determine whether CESM is superior to conventional 2D mammographic screening using a multi-case multi-reader study model.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of malignancy
Groups:
- CESM; Screening 2D Mammography: Recruited patient images were added to other patient images who had both CEM and MRI before biopsy. The images were included in a reader study evaluating diagnostic accuracy of CEM vs 2D MAmmography
Arm/Group | CESM | Screening 2D Mammography
Number analyzed (Participants) | 132 | 132
Probability of malignancy | .906 [.885 to .926] | .788 [.756 to .820]

ADVERSE EVENTS:
Time Frame: Adverse Data were collected at the time of any research imaging exams that were acquired and within 1 year of the exam.
Groups:
- Screening CESM Before Biopsy; Screening MRI Before Biopsy: Each enrolled participant will receive both a CESM and MRI exam prior to the breast biopsy, if they had not been performed already as part of clinical care.
  MRI: Breast MRI will be performed, if not already performed as part of clinical care.
  CESM: After the MRI is complete, patients will be brought to the mammography department for the contrast enhanced mammogram. The CESM will only occur if not already performed as part of the patient's clinical care.
  Biopsy: Patients will then have their biopsy. Any additional findings seen on the CESM or MRI will be worked up also.
  Reader Study: The CESM and the MRI images will be included in a case set that is ready by 10 study radiologists at a later date, after the biopsy is performed. These radiologists will look at the images to see if CESM and MRI find the same number of breast cancers.
  CESM: Contrast enhanced mammography is a new type of mammogram. It uses contrast material combined with the mammogram to highlight areas that might be breast cancer and that could be missed on the mammogram alone
  MRI: MRI uses magnets to create a detailed image of the tissues and bones inside of the body
Arm/Group | Screening CESM Before Biopsy | Screening MRI Before Biopsy
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/132
Other Adverse Events (participants affected / at risk) | 0/132 | 0/132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT03482557/Prot_SAP_002.pdf
  • Informed Consent Form (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03482557/ICF_001.pdf